CLINICAL TRIAL: NCT03210181
Title: Superficial Cervical Plexus Block for Neck and Shoulder Pain Due to Levator Scapulae Syndrome: a Randomized, Double Blind Clinical Trial
Brief Title: Superficial Cervical Plexus Block for Neck and Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Zoher Naja, Chairperson of Anesthesia and Pain Management Department, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1072013
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Neck Pain; Shoulder Pain
MeSH Terms: conditions — Neck Pain; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block (Experimental): Patients will receive superficial cervical plexus block
  Interventions: Other: Superficial cervical plexus block
- Placebo (Placebo Comparator): Patients will receive normal saline
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Superficial cervical plexus block — A nerve stimulator is used to guide the superficial cervical block. The nerve stimulator needle is first passed over the skin after aseptic preparation from the distal to proximal part of the posterior border of the sternocleidomastoid. Upon contraction of the levator scapulae, a mark is placed and the skin is infiltrated with 1 ml lidocaine 1%. A 22-G, 2.5 cm nerve stimulator needle is subsequently advanced through the skin by 0.5-1 cm depending on patient's weight while passing 5-8.5 mA current at 1 Hz. Then, the stimulating current is reduced to 0.5-0.6 mA while maintaining muscle contraction. At this point, 3-5 ml of the anesthetic mixture is injected.
  Arms: Block
Other: Placebo — Patients will receive an equivalent volume of normal saline
  Arms: Placebo

SUMMARY:
Myofascial pain is an important cause of neck pain or neck and shoulder pain. Neck shoulder pain is a common socioeconomic problem that negatively affects the quality of life. Different treatment strategies with limited effectiveness or application have been implemented. However, medication remains a widely used approach.

The levator scapulae is one of the muscles involved in myofascial pain leading to levator scapulae syndrome. The muscle limits the rotation of the neck. It is innervated by branches of the third and fourth cervical nerves through the cervical plexus. Hence, performing superficial cervical plexus block may have some potential effect in reducing myofascial pain.

DETAILED DESCRIPTION:
Patients are randomly divided into two equal groups using the computer-based sealed envelope technique. Group I (Block) will receive superficial cervical plexus block and group II (Placebo) will receive placebo. The physician, patient and data collector are all blind to the patients' assigned group.

Demographic data including gender, age, BMI and American Society of Anesthesiologists (ASA) physical status will be noted at the initial visit. Moreover, patients' medical history, pain history, characteristics and type of pain, as well as previous treatment are collected for each patient. In addition, side effects, pain scores and analgesic consumption will be recorded after performing the block.

Patients will receive 14 daily charts to record daily pain scores, symptoms and the use of analgesics. Patients will be told to take their medications as usual. They will be contacted via phone calls to ensure that they are recording information in the charts.

Pain is assessed using the visual analogue scale (VAS). Patients with score <4 are given 500 mg paracetamol with a maximum of 6 tables per day, or ketoprofen 100 mg tablet to a maximum of 3 tables per 24 hours. Patients with a score>4 are given tramadol hydrochloride 100 mg tablet to a maximum of 3 tablets per day.

Superficial cervical plexus block technique A nerve stimulator is used to guide the superficial cervical block. The nerve stimulator needle is first passed over the skin after aseptic preparation from the distal to proximal part of the posterior border of the sternocleidomastoid. Upon contraction of the levator scapulae, a mark is placed and the skin is infiltrated with 1 ml lidocaine 1%. A 22-G, 2.5 cm nerve stimulator needle is subsequently advanced through the skin by 0.5-1 cm depending on patient's weight while passing 5-8.5 mA current at 1 Hz. Then, the stimulating current is reduced to 0.5-0.6 mA while maintaining muscle contraction. At this point, 3-5 ml of the anesthetic mixture is injected. Each 10 ml of the anesthetic mixture contains: 3ml lidocaine 2%, 3 ml lidocaine 2% with epinephrine 1:200,000, 3 ml bupivacaine 0.5% and 1 ml clonidine 150µg/ml. Group II will receive an equivalent volume of normal saline.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years,
* have neck shoulder pain non-radiating to the arm,
* tenderness in levator scapulae
* refractory to oral analgesics, antiinflammatory medication and physical therapy
* have negative radiographs and bone scans of the shoulders and cervical spine.

Exclusion Criteria:

* organic disease of the brain or spinal cord,
* radiculopathy,
* malignancy,
* hypothyroidism,
* complete blood count (CBC) with high creatine phosphokinase (CPK)
* myopathy,
* autoimmune diseases that are associated with sub clinical myopathy,
* fibromyalgia,
* coagulopathy
* have allergy to bupivacaine,
* taking glucocorticoid and statins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
Analgesic consumption | 2 weeks
  Patients will record the type and amount of analgesics they consume daily

SECONDARY OUTCOMES:
Pain | 2 weeks
  Patients will record their pain using the Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Makassed General Hospital, Beirut, Lebanon